CLINICAL TRIAL: NCT03506217
Title: Hemodynamic Monitorization Using Pulse Counter Vigileo-Flotrac Cardiac Output System in Transapical Off-pump Minimally Invasive Mitral Valve Repair
Brief Title: Using Pulse Counter Vigileo-Flotrac System in Transapical Off-pump Minimally Invasive Mitral Valve Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva Sayhan, Assistant Professor, Sakarya University
Other Study IDs: neocorda
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Mitral Valve Prolapse
Keywords: mitral valve prolaps,; chorda tendinea,; cardiac output
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mitral valve prolaps: Hemodynamic recovery and anesthesia revealed by invasive arterial cardiac output (CO) measurement (Vigileo Flo-trac device) in 13 cases who underwent mitral valve (MV) repair with the transapical off-pump minimally invasive method in our clinic.
  Interventions: Device: Vigileo Flo-trac device

INTERVENTIONS:
Device: Vigileo Flo-trac device — A Vigileo Flotrac pulse counter invasive arterial cardiac output meter was used for cardiac output measurement. Heart rate, blood pressure, cardiac output, stroke volume variance (SVV), systemic vascular resistance (SVR) values were recorded.

SUMMARY:
Minimally invasive transapical off-pump chordae implantation includes features such as tachycardia, arrhythmia, hemorrhage, sudden hemodynamic changes caused by the device moving in the left ventricle and the atrium, for anesthetists. In this observational study, the investigators presented the investigators's hemodynamic recuperation and anesthesia experiences revealed by cardiac output measurement after transapical mitral valve repair.

DETAILED DESCRIPTION:
In Sakarya University Educational Research Hospital, perioperative file records of 13 patients who underwent mitral valve repair using the Neochord DS1000 system were retrospectively analyzed. In addition, hemodynamic measurements recorded with the Vigileo Flotrac invasive arterial cardiac output device were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients that surgical criteria for Neochord implantation with transapical mini-thoracotomy are prolapsus or chordae rupture in posterior, anterior areas or in both leaflets were included.

Exclusion Criteria:

* Exclusion criteria are active endocarditis, functional or ischemic mitral insufficiency (MI), excessive calcific valves, leaflet perforation, anemic dilatation and severe left ventricular dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients who underwent mitral valve repair with Neochord DS1000 system after severe mitral insufficiency in Sakarya University Educational Research Hospital between September-2016 and June-2017
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
invasive arterial cardiac output (CO) measurement | 1 month
  A Vigileo Flotrac pulse counter invasive arterial cardiac output meter was used for cardiac output measurement.
systemic vascular resistance (SVR) | 1mounth
  Systemic vascular resistance is used in calculations of blood pressure, blood flow, and cardiac function. Vasoconstriction (i.e., decrease in blood vessel diameter) increases SVR, whereas vasodilation (increase in diameter) decreases SVR
stroke volume variance (SVV) | 1 mounth
  Stroke volume variation is a naturally occurring phenomenon in which the arterial pulse pressure falls during inspiration and rises during expiration due to changes in intra-thoracic pressure secondary to negative pressure ventilation (spontaneously breathing).
blood pressure | 1 mounth
  The first (or top) number is your systolic blood pressure. It is the highest level your blood pressure reaches when your heart beats. The second (or bottom) number is your diastolic blood pressure. It is the lowest level your blood pressure reaches as your heart relaxes between beats.

CONTACTS AND LOCATIONS:
Overall Officials: Umit Karadeniz, Study Chair — Sakarya University Research and Training Hospital
Locations (1):
- Sakarya University Research and Training Hospital, Sakarya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Colli A, Zucchetta F, Torregrossa G, Manzan E, Bizzotto E, Besola L, Bellu R, Sarais C, Pittarello D, Gerosa G. Transapical off-pump mitral valve repair with Neochord Implantation (TOP-MINI): step-by-step guide. Ann Cardiothorac Surg. 2015 May;4(3):295-7. doi: 10.3978/j.issn.2225-319X.2015.05.01. No abstract available. PMID 26309835